CLINICAL TRIAL: NCT03430011
Title: Protocol H125001: An Open-Label Phase 1/2 Study of JCARH125, BCMA-targeted Chimeric Antigen Receptor (CAR) T Cells, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study Evaluating the Safety and Efficacy of JCARH125 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Acronym: EVOLVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H125001
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: JCARH125; chimeric antigen receptor; multiple myeloma; CAR T cells; B-cell maturation antigen; BCMA; autologous T-cell therapy; immunotherapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JCARH125 (Experimental): Subjects will receive a course of lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by a single dose of JCARH125
  Interventions: Biological: JCARH125
- JCARH125 + anakinra (Experimental): Subjects will receive a course of lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by prophylactic treatment with anakinra and a single dose of JCARH125
  Interventions: Biological: JCARH125 + anakinra

INTERVENTIONS:
Biological: JCARH125 — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCARH125. During JCARH125 production, participants may receive bridging chemotherapy for disease control. Following successful generation of JCARH125 product, participants will receive a course of lymphodepleting chemotherapy followed by one dose of JCARH125 administered intravenously (IV).
  Arms: JCARH125
Biological: JCARH125 + anakinra — Participants will undergo leukapheresis to isolate PBMCs for the production of JCARH125. During JCARH125 production, participants may receive bridging chemotherapy for disease control. Following successful generation of JCARH125 product, participants will receive a course of lymphodepleting chemotherapy followed by two doses of anakinra administered subcutaneously and one dose of JCARH125 administered IV. Subjects receive anakinra for 5 consecutive days following JCARH125 infusion.
  Arms: JCARH125 + anakinra

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study to determine the safety and efficacy of JCARH125, a CAR T-cell product that targets B-cell maturation antigen (BCMA), in adult subjects with relapsed and/or refractory multiple myeloma. The study will include a Phase 1 part to determine the recommended dose of JCARH125 in subjects with relapsed and/or refractory multiple myeloma, followed by a Phase 2 part to further evaluate the safety and efficacy of JCARH125 at the recommended dose. The safety and tolerability of JCARH125 in subjects who receive prophylactic treatment with anakinra will be evaluated in a separate Phase 1 cohort. The antitumor activity of JCARH125 in subjects who have been previously treated with BCMA-directed therapy will be evaluated in separate Phase 2a cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of multiple myeloma (MM) with relapsed and/or refractory (R/R) disease. Participants must have received at least 3 prior anti-myeloma treatment regimens. Participants must have previously received all of the following therapies and must be refractory to the last line of therapy prior to entering the study (not applicable to Phase 2a):

   1. Autologous stem cell transplant
   2. A regimen that included an immunomodulatory agent (eg, thalidomide, lenalidomide, pomalidomide) and a proteasome inhibitor (eg, bortezomib, carfilzomib, ixazomib), either alone or in combination
   3. Anti-CD38 (eg, daratumumab) as part of a combination regimen or as a monotherapy

   Subjects who have received prior allogeneic stem cell transplant or donor lymphocyte infusion at least 100 days before enrollment with no signs of acute or chronic graft-versus-host disease (GVHD) will be considered eligible. Subjects who were not candidates to receive one or more of the above treatments (ie, contraindicated) are eligible.
2. Subjects must have measurable disease.
3. Subject must be willing to provide fresh bone marrow biopsy samples during Screening (and prior to study treatment, if required).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. Adequate renal, bone marrow, hepatic, pulmonary, and cardiac function
6. Phase 2a cohorts only - Subjects with R/R MM who have been previously treated with prior BCMA-directed anti-myeloma therapy, achieved at least a partial response (PR) and progressed on the following treatment:

   1. Subjects who have received prior BCMA-directed CAR T-cell therapy. The last CAR T-cell therapy must have been received at least 6 months prior to JCARH125 screening.
   2. Subjects who have received prior BCMA-directed T-cell engager therapy.
   3. Subjects who have received prior BCMA-directed antibody-drug conjugate therapy.

Exclusion Criteria:

1. Subjects with known active or history of CNS involvement by malignancy
2. Subjects with solitary plasmacytoma; active or history of plasma cell leukemia (PCL); Waldenstrom's macroglobulinemia; Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal plasmaproliferative disorder, Skin changes (POEMS) syndrome; or symptomatic amyloidosis
3. Subjects who are considered eligible to receive and have not refused an autologous stem cell transplant
4. History of another primary malignancy that has not been in remission for at least 3 years. The following are exempt from the 3-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear, and in situ breast cancer that has been completely resected.
5. Require systemic immunosuppressive therapies (eg, calcineurin inhibitors, methotrexate, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-IL-6 or anti-IL-6 receptor [IL-6R])
6. Prior CAR T-cell or other genetically-modified T-cell therapy (not applicable for subjects enrolled in Phase 2a cohorts)
7. Prior treatment with a BCMA-targeted agent (not applicable for subjects enrolled in Phase 2a cohorts)
8. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
9. Untreated or active infection at time of initial screening, at the time of leukapheresis, within 72 hrs before lymphodepletion, or 5 days before JCARH125 infusion.
10. History of any of the following cardiovascular conditions within 6 months of screening: Class III or IV heart failure as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant cardiac disease
11. Subjects with known hypersensitivity to E Coli-derived proteins (only applicable to subjects in Phase 1 Anakinra Cohort)
12. History of severe immediate hypersensitivity reaction to any of the protocol-mandated or recommended agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (20):
  - Local Institution - 0006, Birmingham, Alabama
  - Local Institution - 0007, Duarte, California
  - Local Institution - 0059, Los Angeles, California
  - Local Institution - 0010, San Francisco, California
  - Local Institution - 0060, Denver, Colorado
  - Local Institution - 0042, Atlanta, Georgia
  - Local Institution - 0016, New Lenox, Illinois
  - Local Institution - 0061, Indianapolis, Indiana
  - Local Institution - 0053, Westwood, Kansas
  - Local Institution - 0009, Baltimore, Maryland
  - Local Institution - 0005, Boston, Massachusetts
  - Local Institution - 0062, Detroit, Michigan
  - Local Institution - 0054, Rochester, Minnesota
  - Local Institution - 0038, Hackensack, New Jersey
  - Local Institution - 0013, Buffalo, New York
  - Local Institution - 0001, New York, New York
  - Local Institution - 0058, Portland, Oregon
  - Local Institution - 0023, Seattle, Washington
  - Local Institution - 0018, Seattle, Washington
  - Local Institution - 0055, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 50 x 10^6 Cells: JCARH125 IV at dose level 50 x 10^6 consisting of CD3+CAR+T cells
- Phase 1 150 x 10^6 Cells: JCARH125 IV at dose level 150 x 10^6 consisting of CD3+CAR+T cells
- Phase 1 300 x 10^6 Cells: JCARH125 IV at dose level 300 x 10^6 consisting of CD3+CAR+T cells
- Phase 1 450 x 10^6 Cells: JCARH125 IV at dose level 450 x 10^6 consisting of CD3+CAR+T cells
- Phase 1 600 x 10^6 Cells: JCARH125 IV at dose level 600 x 10^6 consisting of CD3+CAR+T cells
- Phase 1 Anakinra 600 x 10^6 Cells: 2 doses of 100 mg anakinra administered subcutaneously (SC) for 5 consecutive days + JCARH125 IV at dose level 600 x 10^6 consisting of CD3+CAR+T cells
- Phase 2 600 x 10^6 Cells: JCARH125 IV at dose level 600 x 10^6 consisting of CD3+CAR+T cells expansion
- Phase 2a 600 x 10^6 Cells Anti-BCMA: JCARH125 IV at dose level 600 x 10^6 consisting of CD3+CAR+T cells in participants previously treated with BCMA-directed anti-myeloma therapy
Period: Pre-Treatment
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Started (Underwent Leukapheresis) | 15 | 30 | 27 | 22 | 22 | 14 | 25 | 10
Received Lymphodepleting Chemotherapy (LDC) | 15 | 30 | 26 | 21 | 20 | 14 | 24 | 10
Completed (Received JCARH125) | 14 | 30 | 26 | 21 | 20 | 14 | 24 | 10
Not Completed | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Screen Fail | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — No JCARH125 - disease related complications | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant not eligible - other reasons | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: JCARH125 Treatment
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Started (Received JCARH125) | 14 | 30 | 26 | 21 | 20 | 14 | 24 | 10
Completed | 8 | 9 | 7 | 6 | 9 | 6 | 11 | 3
Not Completed | 6 | 21 | 19 | 15 | 11 | 8 | 13 | 7
Not completed — Withdrawal by Subject | 1 | 1 | 5 | 5 | 3 | 4 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 4 | 19 | 10 | 8 | 5 | 3 | 4 | 2
Not completed — Other reasons | 1 | 0 | 4 | 2 | 2 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA | Total
Number analyzed (Participants) | 15 | 30 | 27 | 22 | 22 | 14 | 25 | 10 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 19 | 16 | 15 | 14 | 9 | 17 | 5 | 107
  >=65 years | 3 | 11 | 11 | 7 | 8 | 5 | 8 | 5 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 10 | 9 | 10 | 7 | 8 | 6 | 68
  Male | 10 | 17 | 17 | 13 | 12 | 7 | 17 | 4 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 3 | 2 | 1 | 1 | 0 | 12
  Not Hispanic or Latino | 13 | 25 | 25 | 19 | 20 | 12 | 24 | 7 | 145
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 2 | 3 | 2 | 2 | 1 | 17
  White | 9 | 22 | 23 | 16 | 16 | 9 | 20 | 4 | 119
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 2 | 2 | 3 | 2 | 2 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) in Phase 1
Description: DLT is defined as adverse events (AEs) that occur within 21 days following JCARH125 infusion and meet any of the following criteria:
  * Treatment-emergent Grade ≥3 allergic reactions related to JCARH125;
  * Treatment-emergent Grade 3 seizures, regardless of attribution, that do not resolve to Grade ≤2 within 3 days in participants who have no evidence of central nervous system (CNS) involvement of Multiple Myeloma or other CNS pathology;
  * Treatment-emergent autoimmune toxicity Grade ≥3, regardless of attribution (excluding B-cell aplasia);
  * Treatment-emergent Grade 3 CRS that does not resolve to Grade ≤2 within 72 hours;
  * Any other treatment-emergent Grade 3 AE related to JCARH125 that does not resolve to Grade ≤2 within 7 days;
  * Any treatment-emergent Grade 4 AE related to JCARH125 that does not resolve to Grade ≤2 within 7 days;
  * Treatment-emergent Grade 4 Cytokine Release Syndrome of any duration;
  * Any treatment-emergent Grade 5 toxicity not due to the underlying malignancy
Time Frame: From day 1 to day 22 following JCARH125 infusion (Up to 21 days)
Population: All participants who have either experienced a DLT or were followed for the full DLT evaluation period in phase 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells
Number analyzed (Participants) | 15 | 30 | 27 | 22 | 22
Participants | 0 | 1 | 1 | 3 | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity in Phase 1 and Phase 1 Anakinra
Description: TEAE is defined as an AE that starts any time from initiation of JCARH125 administration through and including 90 days following the JCARH125 infusion graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Any AE occurring after the initiation of another anticancer treatment will not be considered a TEAE. Grade 3=Severe; Grade 4=Life-threatening; and Grade 5=death.
Time Frame: From the time of JCARH125 infusion to 90 days following the infusion (Up to 90 days)
Population: All participants who received at least one infusion of JCARH125 (and at least one dose of anakinra as prophylactic intervention for phase 1 Anakinra) in phase 1 and in phase 1 Anakinra
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 14 | 30 | 26 | 21 | 20 | 14
Participants
  TEAE | 14 | 30 | 26 | 21 | 20 | 14
  Grade 3-5 TEAE | 14 | 30 | 25 | 21 | 20 | 13
  Grade 5 TEAE | 0 | 1 | 1 | 2 | 0 | 0
  JCARH125-Related TEAE | 12 | 26 | 25 | 21 | 20 | 14
  JCARH125-Related Grade 3-5 TEAE | 5 | 10 | 15 | 16 | 16 | 7
  JCARH125-Related Grade 5 TEAE | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities by Severity in Phase 1 and Phase 1 Anakinra
Description: Clinically significant laboratory abnormalities are assessed by investigator and are reported as treatment-emergent adverse event (TEAE). TEAE is defined as an AE that starts any time from initiation of JCARH125 administration through and including 90 days following the JCARH125 infusion graded by Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Any AE occurring after the initiation of another anticancer treatment is not considered a TEAE. Grade 3=Severe; Grade 4=Life-threatening.
Time Frame: From the time of JCARH125 infusion to 90 days following the infusion (Up to 90 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 14 | 30 | 26 | 21 | 20 | 14
Participants
  Neutropenia grade 3 | 4 | 1 | 2 | 1 | 3 | 1
  Neutropenia grade 4 | 10 | 28 | 22 | 20 | 17 | 10
  Anemia grade 3 | 9 | 19 | 16 | 11 | 13 | 10
  Thrombocytopenia grade 3 | 0 | 4 | 3 | 1 | 0 | 4
  Thrombocytopenia grade 4 | 4 | 15 | 11 | 12 | 11 | 5
  Leukopenia grade 3 | 0 | 0 | 2 | 1 | 3 | 0
  Leukopenia grade 4 | 4 | 8 | 12 | 7 | 3 | 4
  Lymphopenia grade 3 | 1 | 2 | 4 | 3 | 1 | 1
  Lymphopenia grade 4 | 0 | 1 | 2 | 0 | 1 | 0
  Febrile neutropenia grade 3 | 1 | 7 | 2 | 0 | 0 | 0
  Febrile neutropenia grade 4 | 0 | 0 | 0 | 1 | 0 | 0
  Haemolysis grade 3 | 0 | 0 | 0 | 0 | 1 | 0
  Hypofibrinogenaemia grade 3 | 0 | 0 | 1 | 0 | 0 | 0
  Hypophosphataemia grade 3 | 1 | 5 | 2 | 6 | 6 | 6
  Hypophosphataemia grade 4 | 0 | 1 | 0 | 0 | 0 | 0
  Hypocalcaemia grade 3 | 0 | 2 | 0 | 1 | 2 | 1
  Hypocalcaemia grade 4 | 0 | 0 | 0 | 1 | 0 | 0
  Hypokalaemia grade 3 | 0 | 3 | 0 | 0 | 1 | 0
  Hyponatraemia grade 3 | 1 | 1 | 2 | 1 | 0 | 2
  Hypomagnesaemia grade 3 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycaemia grade 3 | 0 | 0 | 0 | 2 | 0 | 0
  Hyperglycaemia grade 4 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoalbuminaemia grade 3 | 0 | 1 | 0 | 0 | 1 | 1
  Hypertriglyceridaemia grade 3 | 0 | 1 | 0 | 0 | 0 | 0
  Hypertriglyceridaemia grade 4 | 0 | 1 | 0 | 1 | 0 | 1
  Alanine aminotransferase increased grade 3 | 1 | 0 | 0 | 2 | 1 | 1
  Aspartate aminotransferase increased grade 3 | 0 | 2 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased grade 4 | 1 | 1 | 0 | 2 | 0 | 0
  Blood alkaline phosphatase increased grade 3 | 0 | 0 | 0 | 1 | 0 | 0
  Blood bilirubin increased grade 3 | 0 | 0 | 0 | 0 | 0 | 1
  Serum ferritin increased grade 3 | 0 | 1 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Receiving Prophylactic Anakinra With Grade ≥2 Cytokine Release Syndrome (CRS) in Phase 1 and Phase 1 Anakinra
Description: Number of participants receiving prophylactic anakinra with grade ≥ 2 CRS relative to the number of participants treated at the recommended Phase 2 dose (RP2D) in the Phase 1 dose escalation portion of the trial with grade ≥ 2 CRS. CRS grade is defined by the most severe symptom (excluding fever). Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening
Time Frame: From first infusion to up to aproximately 61 months
Population: All participants who received at least one infusion of JCARH125 (and at least one dose of anakinra as prophylactic intervention for phase 1 Anakinra), at dose level 600 x 10^6 in phase 1 and in phase 1 Anakinra
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 20 | 14
Participants | 11 | 4

5. Primary Outcome: Time to Onset of Grade ≥2 Cytokine Release Syndrome (CRS) in Phase 1 and Phase 1 Anakinra
Description: Time to first onset of Grade ≥2 CRS in participants receiving prophylactic anakinra relative to onset of Grade ≥ 2 CRS in participants treated at the RP2D(s) in the Phase 1 dose escalation portion of the trial. Time to onset is calculated from the latest JCARH125 infusion prior to the first onset of Grade >= 2 CRS. CRS grade is defined by the most severe symptom (excluding fever). Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening
Time Frame: From JCARH125 infusion to the first onset of Grade ≥2 CRS (Up to approximately 61 months)
Population: All participants with grade ≥2 CRS who received at least one infusion of JCARH125 (and at least one dose of anakinra as prophylactic intervention for phase 1 Anakinra) at dose level 600 x 10^6 in phase 1 and in phase 1 Anakinra
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 11 | 4
Days | 2.0 [1 to 3] | 2.0 [2 to 3]

6. Primary Outcome: Number of Participants Receiving Prophylactic Anakinra With no Cytokine Release Syndrome (CRS) Occurring on Days 1-3 in Phase 1 Anakinra
Description: The number of participants receiving prophylactic anakinra with no CRS occurring on study days 1, 2, or 3. CRS grade is defined by the most severe symptom (excluding fever). Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening
Time Frame: Day 1, 2, 3
Population: All participants who received at least one infusion of JCARH125 and at least one dose of anakinra as prophylactic intervention in phase 1 Anakinra
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 14
Participants | 2

7. Primary Outcome: Overall Response Rate (ORR) in Phase 2 and Phase 2a
Description: ORR is defined as stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), according to IMWG criteria. Participants without any reported disease response assessments will be considered non-responders.
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates. When the only method to measure disease is by serum FLC levels, CR can be defined as a normal FLC ratio of 0.26 to 1.65; VGPR=serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein level plus urine M-protein level < 100 mg/24 h; PR=≥ 50% reduction of serum M protein plus reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg/24 h
Time Frame: From the time of the JCARH125 infusion until disease progression, end of study, or the start of another anticancer therapy or stem cell transplant (Up to aproximately 61 months)
Population: All participants who received conforming JCARH125 cell product at the recommended phase 2 dose and have measurable disease at the last disease assessment prior to receiving JCARH125 infusion in phase 2 and in phase 2a
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 24 | 10
Percent of participants | 91.7 [73.0 to 99.0] | 100.0 [69.2 to 100.0]

8. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Cmax is the maximal concentration of JCARH125 CAR T cells in the blood after its infusion as determined by quantitative polymerase chain reaction (qPCR) to detect the JCARH125 transgene.
Time Frame: From JCARH125 infusion through the day 29 visit
Population: All participants who have the necessary PK measurements to provide interpretable results for this specific parameter of interest
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies/UG
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 14 | 30 | 26 | 21 | 20 | 14 | 24 | 10
Copies/UG | 61037.57 (365.26) | 64705.82 (305.31) | 123460.33 (156.23) | 122228.99 (174.22) | 162706.00 (83.19) | 176233.64 (99.44) | 140331.08 (234.07) | 103009.98 (128.25)

9. Secondary Outcome: Time to Maximum Observed Concentration (Tmax)
Description: Tmax is the first study day the maximum observed concetration (Cmax) of JCARH125 CAR T cells in the blood is reached as determined by quantitative polymerase chain reaction (qPCR) to detect the JCARH125 transgene.
Time Frame: From JCARH125 infusion through the day 29 visit
Population: as for outcome 8
Measure: Median (Full Range); unit: Day
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 14 | 30 | 26 | 21 | 20 | 14 | 24 | 10
Day | 13.50 [7.0 to 28.0] | 11.00 [4.0 to 22.0] | 10.00 [3.0 to 21.0] | 10.00 [7.0 to 25.0] | 10.00 [3.0 to 23.0] | 13.50 [7.0 to 28.0] | 9.50 [4.0 to 22.0] | 14.50 [7.0 to 21.0]

10. Secondary Outcome: Area Under the Concertation-Time Curve (AUC) From Time Day 1 to Day 29 [AUC (0-28 Days)]
Description: AUC (0-28) of JCARH125 CAR T cells in the blood as determined by quantitative polymerase chain reaction (qPCR) to detect the JCARH125 transgene.
Time Frame: From JCARH125 infusion through 28 days after the infusion
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*copies/UG
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 13 | 30 | 26 | 20 | 20 | 13 | 23 | 10
Day*copies/UG | 556080.86 (288.83) | 610142.64 (276.50) | 1307054.13 (159.86) | 1390556.32 (188.93) | 1956613.78 (80.39) | 2052280.38 (104.12) | 1427277.29 (226.53) | 1287032.03 (145.22)

11. Secondary Outcome: Number of Participants With Pharmacokinetics Persistence
Description: Pharmacokinetics persistence of JCARH125 CAR T cells in the blood as determined by quantitative polymerase chain reaction (qPCR) over time to detect the JCARH125 transgene. Persistence is defined as a transgene count greater than or equal to the lower limit of detection (LLOD).
Time Frame: Day 29, 60, 90, 180, 270, 365, 545, 730
Population: All participants who have the necessary PK measurements to provide interpretable results for the specific parameters of interest
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 14 | 30 | 26 | 20 | 17 | 14 | 23 | 10
Participants
  Day 29 | 14 | 29 | 26 | 20 | 17 | 14 | 23 | 10
  Day 60: number analyzed (Participants) | 12 | 30 | 25 | 17 | 13 | 13 | 22 | 10
  Day 60 | 9 | 26 | 21 | 16 | 13 | 12 | 21 | 10
  Day 90: number analyzed (Participants) | 13 | 24 | 24 | 19 | 11 | 14 | 21 | 8
  Day 90 | 5 | 16 | 20 | 17 | 9 | 13 | 18 | 7
  Day 180: number analyzed (Participants) | 9 | 18 | 21 | 16 | 13 | 10 | 18 | 7
  Day 180 | 2 | 8 | 14 | 12 | 8 | 9 | 13 | 4
  Day 270: number analyzed (Participants) | 7 | 9 | 14 | 8 | 11 | 10 | 14 | 5
  Day 270 | 1 | 2 | 9 | 2 | 9 | 7 | 8 | 4
  Day 365: number analyzed (Participants) | 7 | 7 | 7 | 10 | 12 | 8 | 14 | 5
  Day 365 | 0 | 1 | 4 | 2 | 6 | 4 | 8 | 3
  Day 545: number analyzed (Participants) | 4 | 2 | 6 | 6 | 8 | 3 | 11 | 3
  Day 545 | 0 | 0 | 4 | 4 | 2 | 3 | 3 | 2
  Day 730: number analyzed (Participants) | 0 | 2 | 4 | 3 | 6 | 3 | 5 | 1
  Day 730 | 0 | 0 | 2 | 2 | 4 | 2 | 1 | 1

12. Secondary Outcome: Overall Response Rate (ORR) in Phase 1 and Phase 1 Anakinra
Description: as for outcome 7
Time Frame: From the time of the JCARH125 infusion until disease progression, end of study, or the start of another anticancer therapy or stem cell transplant (Up to 61 approximately months)
Population: All participants who received conforming JCARH125 cell product at the recommended phase 2 dose (and at least one dose of anakinra as prophylactic intervention for phase 1 Anakinra) and have measurable disease at the last disease assessment prior to receiving JCARH125 infusion in phase 1 and in phase 1 Anakinra
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells
Number analyzed (Participants) | 14 | 30 | 26 | 20 | 20 | 14
Percent of participants | 78.6 [49.2 to 95.3] | 86.7 [69.3 to 96.2] | 96.2 [80.4 to 99.9] | 90.0 [68.3 to 98.8] | 100.0 [83.2 to 100.0] | 100.0 [76.8 to 100.0]

13. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as stringent complete response (sCR) or complete response (CR), according to IMWG criteria. Participants without any reported disease response assessments will be considered non-responders.
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates
Time Frame: as for outcome 7
Population: All participants who received conforming JCARH125 cell product at the recommended phase 2 dose (and at least one dose of anakinra as prophylactic intervention for phase 1 Anakinra) and have measurable disease at the last disease assessment prior to receiving JCARH125 infusion
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 14 | 30 | 26 | 20 | 20 | 14 | 24 | 10
Percent of participants | 42.9 [17.7 to 71.1] | 33.3 [17.3 to 52.8] | 46.2 [26.6 to 66.6] | 45.0 [23.1 to 68.5] | 65.0 [40.8 to 84.6] | 35.7 [12.8 to 64.9] | 54.2 [32.8 to 74.4] | 40.0 [12.2 to 73.8]

14. Secondary Outcome: Duration of Response (DoR) in Phase 2 and 2a
Description: DoR is defined as the time from first response (stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR)) to the earlier date of progressive disease or death due to any cause.
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates; VGPR=serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein level plus urine M-protein level < 100 mg/24 h; PR=≥ 50% reduction of serum M protein plus reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg/24 h.
  Progressive disease is defined as (1) Increase of ≥25% from lowest confirmed response; (2) Appearance of a new lesion(s); (3) ≥50% increase in circulating plasma cells.
Time Frame: From first response to the date of progression or death due to any cause, whichever occurs first (Up to approixmately 61 months)
Population: All participants with sCR, CR, VGPR, or PR who received conforming JCARH125 cell product at the recommended phase 2 dose and have measurable disease at the last disease assessment prior to receiving JCARH125 infusion in phase 2 and in phase 2a
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 22 | 10
Months | 18.2 [2 to 23] | 10.1 [1 to 23]

15. Secondary Outcome: Duration of Complete Response (DoCR) in Phase 2 and 2a
Description: DoCR is defined as the time from first response (stringent complete response (sCR), complete response (CR)) to the earlier date of progressive disease or death due to any cause.
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates.
  Progressive disease is defined as (1) Increase of ≥25% from lowest confirmed response; (2) Appearance of a new lesion(s); (3) ≥50% increase in circulating plasma cells.
Time Frame: as for outcome 14
Population: All participants with sCR or CR who received conforming JCARH125 cell product at the recommended phase 2 dose and have measurable disease at the last disease assessment prior to receiving JCARH125 infusion in phase 2 and in phase 2a
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 13 | 4
Months | 18.2 [0 to 23] | 10.8 [3 to 23]

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity in Phase 2 and Phase 2a
Description: as for outcome 2
Time Frame: From the time of JCARH125 infusion to 90 days following the infusion (Up to 90 days)
Population: All participants who received at least one infusion of JCARH125 in phase 2 and in phase 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 24 | 10
Participants
  TEAE | 24 | 10
  Grade 3-5 TEAE | 23 | 9
  Grade 5 TEAE | 2 | 0
  JCARH125-Related TEAE | 23 | 8
  JCARH125-Related Grade 3-5 TEAE | 16 | 7
  JCARH125-Related Grade 5 TEAE | 1 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities by Severity in Phase 2 and Phase 2a
Description: as for outcome 3
Time Frame: From the time of JCARH125 infusion to 90 days following the infusion (Up to 90 days)
Population: All participants who received at least one infusion of JCARH125 in phase 2 and in phase 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 24 | 10
Participants
  Neutropenia grade 3 | 3 | 1
  Neutropenia grade 4 | 18 | 6
  Anemia grade 3 | 11 | 3
  Thrombocytopenia grade 3 | 3 | 0
  Thrombocytopenia grade 4 | 10 | 3
  Leukopenia grade 3 | 1 | 0
  Leukopenia grade 4 | 8 | 1
  Lymphopenia grade 3 | 1 | 0
  Lymphopenia grade 4 | 3 | 0
  Febrile neutropenia grade 3 | 1 | 0
  Hypophosphataemia grade 3 | 6 | 1
  Hypocalcaemia grade 3 | 3 | 0
  Hypocalcaemia grade 4 | 1 | 0
  Hypokalaemia grade 3 | 2 | 0
  Hyponatraemia grade 3 | 2 | 0
  Hyperglycaemia grade 3 | 2 | 0
  Hypertriglyceridaemia grade 3 | 3 | 0
  Lactic acidosis grade 3 | 1 | 0
  Alanine aminotransferase increased grade 4 | 1 | 0
  Aspartate aminotransferase increased grade 3 | 1 | 0
  Aspartate aminotransferase increased grade 4 | 1 | 0
  Blood fibrinogen decreased grade 3 | 1 | 0
  Blood fibrinogen decreased grade 4 | 1 | 0
  CD4 lymphocytes decreased grade 3 | 1 | 0

18. Secondary Outcome: Overall Survival (OS) in Phase 2 and Phase 2a
Description: OS is defined as the time from the JCARH125 infusion until death due to any cause.
Time Frame: Form date of first infusion to the date of death due to any reason (Up to apprixamtely 61 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 24 | 10
Months | NA [8.71 to NA] — insufficient number of participants with events | NA [7.62 to NA] — insufficient number of participants with events

19. Secondary Outcome: Progression Free Survival (PFS) in Phase 2 and Phase 2a
Description: PFS is defined as the time from JCARH125 infusion until the earliest date of disease progression or death from any cause. Progressive disease (PD) is defined as (1) Increase of ≥25% from lowest confirmed response in one or more of the following: Serum M-protein absolute increase ≥0.5 g/dL; Serum M-protein increase ≥1 g/dL, if the lowest M component was ≥5 g/dL; Urine M protein absolute increase ≥200 mg/24 h; the difference between involved and uninvolved FLC levels absolute increase >10 mg/dL; Bone marrow plasma-cell percentage irrespective of baseline status absolute increase ≥10%. (2) Appearance of a new lesion(s), ≥50% increase from nadir in SPDd of >1 lesion, or ≥50% increase in the longest diameter of a previous lesion >1 cm in short axis. (3) ≥50% increase in circulating plasma cells (minimum of 200 cells μL) if this is the only measure of disease.
Time Frame: Form date of first infusion to the date of disease progression, or death, due to any reason (Up to approximately 61 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 24 | 10
Months | 14.75 [5.85 to 23.82] | 12.25 [3.25 to 17.94]

20. Secondary Outcome: Time to Response (TTR) in Phase 2 and Phase 2a
Description: TTR is defined from JCARH125 infusion to the first document of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates; VGPR=serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein level plus urine M-protein level < 100 mg/24 h; PR=≥ 50% reduction of serum M protein plus reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg/24 h.
  Progressive disease is defined as (1) Increase of ≥25% from lowest confirmed response; (2) Appearance of a new lesion(s); (3) ≥50% increase in circulating plasma cells.
Time Frame: as for outcome 19
Population: as for outcome 14
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 22 | 10
Months | 0.99 [0.9 to 12.5] | 0.97 [0.9 to 2.2]

21. Secondary Outcome: Time to Complete Response (TTCR) in Phase 2 and Phase 2a
Description: TTCR is defined from JCARH125 infusion to the first document of stringent complete response (sCR) or complete response (CR).
  sCR=complete response plus normal free light chain ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates.
  Progressive disease is defined as (1) Increase of ≥25% from lowest confirmed response; (2) Appearance of a new lesion(s); (3) ≥50% increase in circulating plasma cells.
Time Frame: as for outcome 19
Population: as for outcome 15
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
Number analyzed (Participants) | 13 | 4
Months | 2.79 [1.0 to 15.2] | 1.41 [1.0 to 2.2]

22. Secondary Outcome: Change From Baseline in the Total Score of European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ-C30) in Phase 2
Description: The EORTC QLQ-C30 is a 30-item scale composed of both multi-item scales and single-item measures such as functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Subscale scores are transformed to 0 to 100 scale, with higher scores on functional scales indicating better function and higher score on symptom scales indicating worse symptoms. Baseline is defined as the last non-missing measurement prior to JCARH125 infusion.
Time Frame: Baseline and visit 24 month
Population: All participants who received at least one infusion of JCARH125 with baseline and post-baseline assessment at the respective visit in phase 2 only as prespecified in the protocol
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Phase 2 600 x 10^6 Cells
Number analyzed (Participants) | 4
Score on a Scale
  Global Health Status/QoL Month 24 | -2.08 (10.49)
  Physical Functioning Month 24 | -6.67 (9.43)
  Role Functioning Month 24 | 0.00 (13.61)
  Emotional Functioning Month 24 | -6.25 (7.98)
  Cognitive Functioning Month 24 | 4.17 (8.33)
  Social Functioning Month 24 | 16.67 (13.61)
  Fatigue Month 24 | 5.56 (6.42)
  Pain Month 24 | -4.17 (8.33)
  Nausea and Vomiting Month 24 | 4.17 (8.33)
  Dyspnea Month 24 | -8.33 (16.67)
  Insomnia Month 24 | 0.00 (27.22)
  Appetite Loss Month 24 | 8.33 (16.67)
  Constipation Month 24 | 8.33 (16.67)
  Diarrhea Month 24 | 8.33 (16.67)
  Financial Difficulties Month 24 | 8.33 (16.67)

23. Secondary Outcome: Change From Baseline in the Total Score of European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (QLQ-MY20) in Phase 2
Description: QLQ-MY20 includes 20 questions across four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score for the disease symptoms scale = higher level of symptomatology.
Time Frame: Baseline and visit 24 month
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Phase 2 600 x 10^6 Cells
Number analyzed (Participants) | 4
Score on a Scale
  Disease Symptoms | 0.00 (0.00)
  Side Effects of Treatment | 6.11 (3.98)
  Future Perspectives | 11.11 (9.07)
  Body Image | 16.67 (33.33)

24. Secondary Outcome: Change From Baseline (EQ-5D-5L) Index Score in Phase 2
Description: EQ-5D-5L is a standardized measure of health status that consists of descriptive system and Visual Analogue scale VAS). The descriptive system comprises dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the dimensions are combined in a 5-digit number corresponding to response categories for successive dimensions using a scoring algorithm. The VAS system has endpoints labeled "the best health you can imagine" and "the worst health you can imagine." The scale is numbered from 0 to 100 with 0 corresponding to the worst imaginable health state and 100 corresponding to the best imaginable health state. A high score represents a better level of quality of life
Time Frame: Baseline and visit 24 month
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 600 x 10^6 Cells
Number analyzed (Participants) | 4
Score on a scale
  Mobility Index Score | -0.3 (0.5)
  Self Care Index Score | 0.0 (0.0)
  Activity Index Score | 0.3 (0.5)
  Pain Index Score | 0.0 (0.0)
  Anxiety Index Score | 0.3 (1.0)
  Utility Index US Index Score | -0.0035 (0.1193)

25. Secondary Outcome: Duration of Hospitalization From JCARH125 Administration in Phase 2
Description: Total length of all intensive care unit (ICU) and non-ICU stays from JCARH125 Administration. ICU inpatient and non-ICU inpatient are not exclusive. Total length includes participants who had multiple hospitalization stays.
Time Frame: From JCARH125 infusion to up to approximately 61 months
Population: as for outcome 22
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 2 600 x 10^6 Cells
Number analyzed (Participants) | 24
Days
  ICU inpatient: number analyzed (Participants) | 9
  ICU inpatient | 9.0 [3 to 32]
  non-ICU inpatient: number analyzed (Participants) | 21
  non-ICU inpatient | 11.0 [6 to 58]

26. Secondary Outcome: Reasons for Hospitalization From JCARH125 Administration in Phase 2
Description: Number of participants with reasons for hospitalization from JCARH125 administration
Time Frame: From JCARH125 infusion to up to approximately 61 months
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 600 x 10^6 Cells
Number analyzed (Participants) | 24
Participants
  Adverse Event | 3
  Prophylaxis | 21

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from the first participant undergoing leukapheresis until their study completion (up to approximately 61 months). SAEs and other AEs were assessed from first JCARH125 infusion until 90 days following the JCARH125 infusion (up to approximately 41 months).
Description: The total number at risk for all-cause mortality represents all participants who underwent leukapheresis. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants that received at least 1 infusion of study medication (JCARH125).
Arm/Group | Phase 1 50 x 10^6 Cells | Phase 1 150 x 10^6 Cells | Phase 1 300 x 10^6 Cells | Phase 1 450 x 10^6 Cells | Phase 1 600 x 10^6 Cells | Phase 1 Anakinra 600 x 10^6 Cells | Phase 2 600 x 10^6 Cells | Phase 2a 600 x 10^6 Cells Anti-BCMA
All-Cause Mortality (participants affected / at risk) | 5/15 | 22/30 | 14/27 | 9/22 | 7/22 | 4/14 | 6/25 | 2/10
Serious Adverse Events (participants affected / at risk) | 1/14 | 14/30 | 7/26 | 7/21 | 7/20 | 5/14 | 11/24 | 1/10
Other Adverse Events (participants affected / at risk) | 14/14 | 30/30 | 26/26 | 21/21 | 20/20 | 14/14 | 24/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 50 x 10^6 Cells (N=14) | Phase 1 150 x 10^6 Cells (N=30) | Phase 1 300 x 10^6 Cells (N=26) | Phase 1 450 x 10^6 Cells (N=21) | Phase 1 600 x 10^6 Cells (N=20) | Phase 1 Anakinra 600 x 10^6 Cells (N=14) | Phase 2 600 x 10^6 Cells (N=24) | Phase 2a 600 x 10^6 Cells Anti-BCMA (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 3 | 2 | 2 | 2 | 3 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cystitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 50 x 10^6 Cells (N=14) | Phase 1 150 x 10^6 Cells (N=30) | Phase 1 300 x 10^6 Cells (N=26) | Phase 1 450 x 10^6 Cells (N=21) | Phase 1 600 x 10^6 Cells (N=20) | Phase 1 Anakinra 600 x 10^6 Cells (N=14) | Phase 2 600 x 10^6 Cells (N=24) | Phase 2a 600 x 10^6 Cells Anti-BCMA (N=10)
Anaemia (Blood and lymphatic system disorders) | 9 | 21 | 17 | 13 | 15 | 11 | 18 | 5
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 1 | 1 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 8 | 14 | 9 | 6 | 5 | 9 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 6 | 3 | 2 | 1 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 14 | 29 | 24 | 21 | 20 | 11 | 21 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 21 | 16 | 14 | 14 | 9 | 19 | 4
Bradycardia (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 3 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 3 | 1 | 2 | 1 | 1 | 3 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 2 | 4 | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 5 | 8 | 7 | 3 | 6 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 13 | 5 | 5 | 3 | 6 | 8 | 2
Vomiting (Gastrointestinal disorders) | 2 | 6 | 3 | 6 | 2 | 1 | 5 | 0
Asthenia (General disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 3 | 0
Catheter site dermatitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 3
Fatigue (General disorders) | 4 | 9 | 5 | 6 | 5 | 5 | 8 | 3
Gait disturbance (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 8 | 4 | 6 | 3 | 1 | 4 | 2
Pain (General disorders) | 0 | 1 | 0 | 4 | 1 | 0 | 3 | 1
Pyrexia (General disorders) | 5 | 5 | 3 | 2 | 1 | 5 | 5 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 9 | 21 | 21 | 19 | 16 | 11 | 19 | 7
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 4 | 4 | 2 | 0 | 4 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 2 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 4 | 0 | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 1 | 3 | 1 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 0 | 5 | 6 | 3 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 1 | 5 | 4 | 4 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 1 | 3 | 1 | 2 | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Enterovirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 0
Serum ferritin increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 7 | 6 | 5 | 2 | 5 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 2 | 4 | 4 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 3 | 6 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 5 | 5 | 4 | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 14 | 5 | 6 | 6 | 4 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 9 | 2 | 4 | 5 | 4 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 3 | 2 | 6 | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 9 | 7 | 7 | 9 | 7 | 8 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 4 | 3 | 4 | 3 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2 | 2 | 2 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 1
Cognitive disorder (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 4 | 1 | 3 | 2 | 3 | 0
Dysaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 8 | 8 | 8 | 4 | 4 | 6 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 2 | 2 | 3 | 1 | 4 | 0
Depression (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 5 | 4 | 0 | 3 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 2 | 2 | 2 | 0 | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 2 | 0 | 0 | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 5 | 1 | 3 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 5 | 2 | 0 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1 | 2 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 2 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 3 | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 6 | 2 | 2 | 3 | 0 | 4 | 0
Hypotension (Vascular disorders) | 3 | 4 | 4 | 3 | 5 | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03430011/Prot_SAP_000.pdf